CLINICAL TRIAL: NCT01478906
Title: To Investigate Difference of Plasma Orexin A Levels Between Elderly and Youth Patients at Emergence From Sevoflurane-fentanyl Anesthesia Undergoing Elective Lumbar Surgery
Brief Title: Difference of Plasma Orexin A Levels Between Elderly and Young Patients at Emergence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: mzk2010orexin
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Anesthesia

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- elderly ,adult

SUMMARY:
The current study is designed to investigate the difference of plasma orexin A levels between elderly and young patients at emergence from sevoflurane-fentanyl anesthesia who will undergo elective lumbar surgery.

DETAILED DESCRIPTION:
BACKGROUND:A specific group of neurons in the brain produces hypocretin, also called orexin, a peptide which has been established as an important regulator of anesthesia and emergence in the latest few years. In the animal experiment,we found that the level of orexin A in aged rats was higher when compared with that of the young ones. Whereas the numbers of both the orexin receptor 1 and 2 in aged rats decreased. We wonder if there is a similar phenomenon in human beings which might account for the difference between the intervals of elderly and young patients recovering from anesthesia. This study aims to investigate difference of plasma orexin A levels between elderly patients and young at emergence from sevoflurane-fentanyl anesthesia.

DESIGNING:Forty patients with ASA physical status I or II scheduled for elective lumbar surgery under general anesthesia (lasting for 2h to 4h)were enrolled. Anesthesia was induced with propofol 1-1.5mg/kg and fentanyl 2-3μg/kg. Following muscle relaxation with iv rocuronium bromide 1mg/kg endotracheal intubation was performed. Anesthesia was maintained with sevoflurane(inhalational concentration: 0.8-1.5 MAC) fentanyl (total 6μg/kg) and target controlled infusion remifentanil (targeted concentration:2-7ng/ml ) along with an oxygen/air mixture (FiO2 = 0.5). Muscle relaxation was maintained with intermittent rocuronium. Inhalational concentration of sevoflurane and injected target concentration were titrated to maintain the bispectral index (BIS) between 45 and 65 during anesthesia. The end-tidal carbon dioxide level was maintained between 30 and 40mmHg by controlled mechanical ventilation. When the surgery was complicated we adjust the concentration sevoflurane to 0.8MAC of the patient and targeted concentration of remifentanil to 2ng/ml and then stop all anesthetics . Record time from stopping anesthetics to emergence. Arterial blood (2ml) was collected at the following time, such as before and 1h after induction of anesthesia, at emergence (1min after tracheal extubation) and half an hour after tracheal extubation. This was centrifuged at 3000 rpm for 15min at -4 ◦C in order to separate plasma then stored at -80 ◦C until assay for orexin A concentrations.

EXPECTED RESULTS:The plasma orexin A of group elderly will be higher with the emergence time longer than youth patients.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is Adult (≥18 years old )
2. Participants with a Body Mass Index (BMI) 20-25 kg/m2 at the prestudy (screening) visit.
3. Participants with ASA physical status Ⅰor Ⅱ
4. Participants with Heart function rating Ⅰor Ⅱ
5. Glucose of patients is lower than 8 mmol/L
6. patients will undergo elective lumbar surgery

Exclusion Criteria:

1. Participant is a pregnant woman or a nursing mother.
2. Participants have a history of narcotics allergic reactions
3. indices of liver or kidney function is twice higher than normal
4. Participants have a history or diagnosis of depression
5. Participants have a history of Brain Trauma
6. Participants have a history of narcotics addiction or drug addiction
7. Participants have a history or diagnosis of adrenal gland diseases
8. Participants or his family have an International Classification of Sleep Disorders diagnosis of OSA

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 to 80 years old ,undergo Lumbar Surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-06 (Estimated); Study Completion 2012-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hailong Dong, MD,PhD, Study Director — Xijing Hospital
Locations (1):
- Anesthesiology department of Xijing Hospital, Xi'an, Shaanxi, China